CLINICAL TRIAL: NCT05660460
Title: A Study of the Incidence and Treatment of Impaired Lung Function Among Socially Vulnerable Individuals at a Street Level
Brief Title: COPD at a Street Level
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Brugernes Akademi (Unknown)
Responsible Party: Principal Investigator, Charlotte Suppli Ulrik, Professor, consultant, Hvidovre University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: H-22046465
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: COPD
Keywords: screening; socially vulnerable patients; mobile clinic
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Spirometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Socially vulnerable individuals in contact with a mobile clinic (Other): After obtaining informed consent, a project nurse in the mobile clinic reviews the online-questionnaire with the participant and performs a lung function examination requiring the individual to blow into a plastic tube. If the participant is identified as having obstructive reduction of lung function, they are offered a referral and patient support to a local pulmonary medicine department or GP for further investigation - regardless of whether or not they have a diagnosed or undiagnosed lung disease. In addition, participants are questioned about their motivation for smoking cessation and are informed of the options for this (in hospital and/or referral to the municipality).
  Interventions: Diagnostic Test: Spirometry

INTERVENTIONS:
Diagnostic Test: Spirometry — The method of examination, Spirometry, is noninvasive (i.e. not an intervention that involves penetration into the body by means of incisions or injections.). It is a routine examination and there are no risks, adverse reactions, or discomforts associated with the examination.

SUMMARY:
The trial investigates and describes the prevalence of COPD among socially vulnerable individuals who come in contact with a mobile clinic and investigates the effect of opportunistic screening for COPD in these vulnerable persons. The study population is individuals who come in contact with a mobile clinic, that visits home shelters, open drugs scenes etc. in the Capital Region of Denmark during the inclusion period, and monitor them for up to 1 year in order to investigate variables that are significant in terms of the patients' treatment, hospitalizations, and mortality in relation to COPD. Our hypothesis is that there will be a higher incidence of COPD among socially vulnerable individuals who come in contact with the mobile clinic than in the general population.

DETAILED DESCRIPTION:
The study consists of three sub-studies: A. a descriptive cross-sectional study "The prevalence of COPD among socially vulnerable individuals who come in contact with a mobile clinic" followed by study B a cohort study "The effect of opportunistic screening for COPD among socially vulnerable individuals who come in contact with a mobile clinic", based on a closed cohort, and study C "A qualitative study of patient experiences with screening and treatment of COPD.

People in the lower social classes are at increased risk of developing COPD due to their lifelong accumulation of risk factors, such as smoking, passive smoking and the influence of lifestyle and the environment. In the group with the socially vulnerable individuals, 70% are smokers compared to 18% in the general Danish population. The socially vulnerable individuals are defined here as people affected by homelessness, drug abuse, harmful alcohol consumption, mental illness and poverty. Despite the socially vulnerable group having an over-consumption of general practice visits, 25% of socially vulnerable individuals state that they do not have contact with or use their own doctor. Our hypothesis is therefore that there will be a higher incidence of COPD among socially vulnerable persons who come in contact with the mobile clinic. Purpose: To investigate and describe the prevalence of COPD among socially vulnerable individuals who come in contact with a mobile clinic and to investigate the effect of opportunistic screening for COPD in these vulnerable citizens, followed by a qualitative study of patient experiences with COPD treatment.

Data collection:

Baseline data from the cross-sectional study are derived from lung function measurement and REDCap online-questionnaires completed on inclusion. The data from the cohort study regarding disease burden and hospital visits originates from the national patient registry (LPR) and mortality data is retrieved from the Danish Register of Causes of Death. Data regarding redeemed prescriptions for COPD medicine originates from the Prescription Database. The patients' connection to the job market and income status are based on extracts from RAS (Registry-based Labour Force Statistics), which is administered by Statistics Denmark. Data regarding the highest acquired education (HFAUDD) is from Statistics Denmark.

Variables:

There will be collected the following variables at inclusion: information on demographics, lung function, selv-reported information on: risk factors, socioeconomic variables and symptoms of lung disease. Moreover register data on socioeconomic status, morbidity, physical health by Charlson score, mortality, hospital visits and prescriptions for COPD Medicine will be retrieved after a 1 year follow-up.

Sample size:

To detect a difference between the patient group and the Danish population of minimum 100% a total of 511 participants are needed in the study (power of 80%, p-values=0,05, an estimated COPD prevalence of 4,3% in the Danish population). The collected data will be kept in accordance to the Data Protection Agency guidelines. The studies are carried out in accordance with the principles of the Helsinki Declaration.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Able to speak and understand Danish or English to such an extent that informed consent can be obtained

Exclusion Criteria:

- Not having a Danish civil registration number, since foreign patients do not have free access to examinations and medical treatment, and cannot be followed up in the national patient registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 511 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2027-03-15 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of COPD | Baseline
  1. Prevalence of obstructive lung function reduction among socially vulnerable
Undiagnosed COPD | Baseline
  2. Prevalence of previously undetected COPD
Adherence to first appointment | Baseline
  3. Numbers of socially vulnerable individuals diagnosed with obstructive lung function that are subsequently examined at a pulmonary medicine outpatient clinic/GP
Subscription at first appointment | Baseline
  4. Number of socially vulnerable individuals who after COPD diagnosis are subscribed medical treatment

SECONDARY OUTCOMES:
Smoking status | Baseline
  5. Prevalence of socially vulnerable individuals who smoke and wish to stop smoking
COPD and smoking cessation | Baseline
  6. Prevalence of socially vulnerable individuals with impaired lung function who have a desire to stop smoking
smoking cessation invitation | Baseline
  7. Prevalence of socially vulnerable individuals who want to quit smoking and accept the smoking cessation offers
Adherence to treatment | Baseline
  8. Prevalence of socially vulnerable individuals who claim their prescription for COPD medication
Health service barriers | Baseline
  9. Patient-perceived barriers with COPD treatment through outpatient clinic/GP

CONTACTS AND LOCATIONS:
Overall Officials: Jannet van der Veen, Study Chair — Brugernes Akademi; Charlotte S Ulrik, Principal Investigator — Amager and Hvidovre Hospital
Locations (1):
- Brugernes Akademi, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No